CLINICAL TRIAL: NCT03254979
Title: How to Engage Primary Health Care Providers in an Inter-professional Collaborative Modeling Process for the Optimization of Type-2 Diabetes Primary Prevention: a Randomized Hybrid Implementation Trial
Brief Title: Optimizing the Primary Prevention of Type-2 Diabetes in Primary Health Care
Acronym: PREDIAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Alvaro Sanchez Perez, PhD, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PI15/00350
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Interprofessional Relations; Primary Health Care/Organization & Administration; Diabetes Mellitus, Type 2/Prevention & Control; Primary Prevention/Methods; Risk Reduction Behavior; Randomized Controlled Trial; Life Style
MeSH Terms: conditions — Diabetes Mellitus; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: The implementation strategy to facilitate the adoption of the recommended clinical intervention in primary prevention of T2DM will be common to both comparison groups. In order to differentiate and isolate the effect of the procedure of creation of the Multi-professional Community of Practice, the centers have been randomly assigned to two comparison groups: 5 centers assigned to the sequential procedure and the other 4 centers to the group procedure.
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the new program is an optimization of the type-2 diabetes prevention services already offered in Osakidetza, it is expected that the participating patients will be blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential engagement (Experimental): Inter-professional collaborative practice directed by a local leader and an external facilitator to optimize the integration of a T2D primary prevention recommended clinical intervention. In this group, a sequential engagement of professional categories, initiated in nursing, which finally involves the whole professional groups of the center (eg. physicians, etc), will be followed
  Interventions: Behavioral: Healthy lifestyle prescription
- Global engagement (Active Comparator): Inter-professional collaborative practice directed by a local leader and an external facilitator to optimize the integration of a T2D primary prevention recommended clinical intervention. In this group, a global strategy of engagement with the participation of all professionals from the beginning, will be followed
  Interventions: Behavioral: Healthy lifestyle prescription

INTERVENTIONS:
Behavioral: Healthy lifestyle prescription — 3 actions for the prevention of DM2 in the clinical setting are recommended:
  1. A screening strategy for people with impaired glucose regulation or high risk of developing DM2, with the following recommendations: screening for DM2 within the strategy of opportunistic screening for CV risk factors in population ≥45 years Or ≥30 years in the presence of a previous risk factor (eg, hypertension); Screening for DM2 based on the presence of a BMI ≥25 in the population aged 40-70 years; Or, risk screening for DM2-FINDRISC in a population of 45-70 years.
  2. With those identified at high risk, perform a structured program of intensive intervention focused on the prescription of personalized plans on lifestyle modification (low calorie and low fat diet, and at least 150 minutes of physical exercise per week).
  3. A follow-up intervention component to maintain the motivation of those interviewed, with more frequent contacts initially, with at least annual review visits.

SUMMARY:
RATIONALE The translation into clinical practice of Primary Care (PHC) of effective and sustainable interventions to prevent of type-2 diabetes (T2D) remains an unresolved challenge. Leadership, active involvement of professionals, facilitation and adaptation to the local context and their determinants are known to be key components in the success of implementation strategies that seek to optimize clinical practice. However, one of the areas in which there is still no evidence is related to the effectiveness of different strategies to engage healthcare professionals in such innovation processes. Especially in real-world Primary Care clinical contexts characterized by work overload and limited time, with marked differentiation of professional status, both at the level of identity and competency.

OBJECTIVES To assess the effect of PHC providers engagement procedure in the creation and execution of a facilitated collaborative modelling process, in the adoption, reach, implementation and effectiveness of the recommended clinical practice for the prevention of type-2 Diabetes

METHODOLOGY

Randomized cluster hybrid trial in which 9 PHC centres from Osakidetza will be allocated to two different strategies to engage professionals and create an inter-professional collaborative practice directed by a local leader and an external facilitator, to optimize the integration of a T2D primary prevention program:

* A strategy focused on the sequential activation: started in nursing, which finally manages to involve the whole center
* A global strategy with the participation of all professionals from the beginning

All centres and PHC professionals will receive training on current guidelines and scientific evidence in primary prevention of T2D and effective interventions to promote healthy lifestyles. Headed by a local leader and an external facilitator, centres will conduct a collaborative structured process to model and adapt the intervention and its implementation to the specific context of professionals and centres, and the determinants of T2D prevention practice. One of the groups will perform this strategy globally, promoting the cooperation of all health professionals from the beginning. The other will perform it sequentially, centred first in nursing, who will lately seek the pragmatic cooperation of physicians and other professionals.

All patients without diabetes aged ≥30 years old who attend at least once in collaborating centres at high risk of developing T2DM (FINDRISC> = 14 points and / or intermediate hyperglycaemia) will be eligible for program inclusion. The main outcome measures focus on observed changes in T2DM prevention clinical practice at centre level after 12 and 24 months, as a result of the implementation of one or another engagement strategy. Secondary outcomes will compare their clinical effectiveness in changing exposed eligible patients' main cardio-metabolic risk factors (Weight, BMI, Cholesterol, Glucose, Triglycerides) and lifestyles behaviours (physical activity and diet) after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients without diabetes aged ≥30 years old who attend at least once in collaborating centres at high risk of developing T2DM (Body Mass Index >=25 or intermediate hyperglycaemia) will be eligible for program inclusion.

Exclusion Criteria:

-

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Implementation of the recommended clinical intervention by health care porfessionals | 12 months
  The proportion of non-diabetic patients at high risk of developing DM2 exposed to the recommended intervention actions : assessing habits, personalized advice, prescription of lifestyle change plans and follow-up

SECONDARY OUTCOMES:
Lifestyle change at patient level | 12 months
  Proportion of exposed patients who change their habits (physical activity and diet) and lose 5% of their body weight

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research Unit of Bizkaia, OSAKIDETZA, Bilbao, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez A, Pablo S, Garcia-Alvarez A, Dominguez S, Grandes G; PREDIAPS Group. Effectiveness of two procedures for deploying a facilitated collaborative modeling implementation strategy-the PVS-PREDIAPS strategy-to optimize type 2 diabetes prevention in primary care: the PREDIAPS cluster randomized hybrid type II implementation trial. Implement Sci. 2021 May 27;16(1):58. doi: 10.1186/s13012-021-01127-x. PMID 34044869
- [Derived] Sanchez A, Rogers HL, Pablo S, Garcia E, Rodriguez I, Flores MA, Galarza O, Gaztanaga AB, Martinez PA, Alberdi E, Resines E, Llarena AI, Grandes G; PREDIAPS Group. Fidelity evaluation of the compared procedures for conducting the PVS-PREDIAPS implementation strategy to optimize diabetes prevention in primary care. BMC Fam Pract. 2021 Feb 11;22(1):34. doi: 10.1186/s12875-021-01378-z. PMID 33573600
- [Derived] Sanchez A, Grandes G, Pablo S, Espinosa M, Torres A, Garcia-Alvarez A; PREDIAPS Group. Engaging primary care professionals in collaborative processes for optimising type 2 diabetes prevention practice: the PREDIAPS cluster randomised type II hybrid implementation trial. Implement Sci. 2018 Jul 11;13(1):94. doi: 10.1186/s13012-018-0783-0. PMID 29996928